CLINICAL TRIAL: NCT02640729
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Cross-over Study of Nelotanserin Versus Placebo in Lewy Body Dementia (LBD) Subjects Experiencing Visual Hallucinations (VH)
Brief Title: Study Evaluating Nelotanserin for Treatment of Visual Hallucinations in Subjects With Lewy Body Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-102-2001
Record Dates: First submitted 2015-12-19; First posted 2015-12-29 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Lewy Body Dementia; Visual Hallucinations
Keywords: Lewy body dementia; Dementia with Lewy bodies; Parkinson's disease dementia; Lewy bodies; Visual hallucinations
MeSH Terms: conditions — Lewy Body Disease; Hallucinations | interventions — nelotanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Nelotanserin (Experimental): Nelotanserin 40mg then nelotanserin 80 mg
  Interventions: Drug: Nelotanserin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nelotanserin — once daily, oral, 20-mg tablets
  Arms: Nelotanserin
Drug: Placebo — once daily, oral, matching tablets
  Arms: Placebo

SUMMARY:
This study seeks to evaluate safety and efficacy of Nelotanserin for the treatment of visual hallucinations in subjects with Lewy body dementia.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, cross-over study in subjects with Lewy body dementia who experience frequent visual hallucinations.

Subjects who meet the randomization criteria enter the double-blind treatment period.

Each subject will be randomized 1:1 to one of the 2 treatment sequences: Nelotanserin in the first treatment period followed by placebo in the second treatment period, or placebo in the first treatment period followed by Nelotanserin in the second treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects at least 50 years of age, with a diagnosis of LBD based on DSM-5 diagnostic criteria or diagnosis of Parkinson's disease dementia (PDD) based on DSM-5 diagnostic criteria;
* Presence of frequent visual hallucinations
* Mini Mental State Examination score ≥ 18

Exclusion Criteria:

* Subjects have a current diagnosis of significant psychotic disorders including, but not limited to, schizophrenia or bipolar disorder
* Subjects' psychotic symptoms are secondary to or better accounted for by another medical condition, psychiatric disorder, or substance abuse
* Subjects with a current serious and/or unstable cardiovascular, respiratory, thyroid, gastrointestinal, renal, hematologic or other medical disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated based on incidence of adverse events (AEs) and significant changes in physical examinations, vital signs, ECGs, and routine clinical laboratory assessments from baseline to the end of each treatment period (28 days). | 28 days
Extrapyramidal signs are assessed with the motor subsection of the Unified Parkinson's Disease Rating Scale (UPDRS, Parts II and III). | 28 days

SECONDARY OUTCOMES:
Change in the frequency and severity of visual hallucinations from baseline to the end of each treatment period (28 days) with Nelotanserin or placebo, as recorded and documented by the patient's caregiver | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Director — Axovant Sciences, Inc., Clinical Research
Locations (10):
- United States (10):
  - US123, Fountain Valley, California
  - US114, Boca Raton, Florida
  - US113, Orlando, Florida
  - US132, Lenexa, Kansas
  - US103, Rochester, Minnesota
  - US129, Lincoln, Nebraska
  - US101, Chapel Hill, North Carolina
  - US104, Cleveland, Ohio
  - US105, Columbus, Ohio
  - US131, San Antonio, Texas